CLINICAL TRIAL: NCT02095457
Title: A Randomized Trial of Routine Computerized Outcome and Process Clinical Measures Monitoring in Mental Health Outpatient Services: Preparing for the Planned Public Mental Health Reform in Israel
Brief Title: Routine Outcome Monitoring in Mental Health Outpatient
Acronym: ROM-Shalvata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Ori Ganor, Ori Ganor, MD, Shalvata Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIHP-R-161-2013; R-161-2013 (Other Grant/Funding Number: The Israel National Institute for Health Policy Research)
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Affective Disorders; Anxiety Disorders; Psychotic Disorders; Personality Disorders
Keywords: Routine Outcome Monitoring; Psychotherapy; Alliance; Feedback Informed Treatment; Mental Health Outpatients
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Psychotic Disorders; Personality Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Frequent Monitoring and Feedback (Active Comparator): In the intervention arm, patients routinely fill short monitoring questionnaires, the results of which are fed back to their therapists and staff. The frequency of monitoring is between once a week to once every three months, depending on the type of therapy
  Interventions: Behavioral: Frequent monitoring and feedback
- Infrequent monitoring without feedback (Sham Comparator): In the control arm, patients will infrequently fill short monitoring questionnaires, the results of which are not fed back to their therapists and staff. The frequency of monitoring is between about once a year
  Interventions: Behavioral: Frequent monitoring and feedback

INTERVENTIONS:
Behavioral: Frequent monitoring and feedback — In the intervention arm, patients routinely fill short monitoring questionnaires, the results of which are fed back to their therapists and staff. The frequency of monitoring is between once a week to once every three months, depending on the type of therapy

SUMMARY:
Scientific Background: Inherent gaps exist between the worlds of research and clinical therapy, especially in mental-health systems. Developed as an important strategy aimed to bridge them, widening efforts worldwide have implemented Routine Outcome Monitoring (ROM), a method devised for systematic ongoing quantitative measurements used in diverse clinical practices, from psychotherapies to psychiatric management. The efficacy of this approach has been repeatedly demonstrated in various measures, such as satisfaction with treatment by patients and therapists, lower drop-out rates, symptomatic benefits, and more.

Objectives: The aim of the current study is to test the feasibility and the clinical benefits of implementation of a Routine Outcome Monitoring System in a public clinical center, as a pioneering project in Israel, at the "Shalvata" Mental Health Center.

Working Hypotheses: Incorporation of a ROM system in routine clinical practice is hypothesized to improve patients' and therapists' overall satisfaction, allow for early detection and intervention in therapeutic raptures, decrease drop-out rates, and improve various clinical outcome measures.

Methods: The suggested study is a two-stage (implementation and intervention) open trial. 900 new outpatients in 'Shalvata' clinics will be recruited and randomized to intervention (ROM) and control groups. Assessment questionnaires will be filled periodically using 'CORE-NET', a computerized system enabling repeated measurements and feedback in a user-friendly and efficient manner.

Data Analysis: The evaluation of the differential influence of monitoring processes on overall efficiency as compared to control group will be tested using Multiple Analysis of Variance (MANOVA). The predictive value of possible variables on process and outcome of therapy will be assessed using stratified regression analyses. The possible causal effects between specific lagged variables will be assessed using Hierarchical Linear Modeling and Time Series Analysis.

Contribution: This pioneering study is the first in Israel to offer a routine systematic evaluation of therapeutic processes, as well as assessing its clinical effects. Consequently, a large and meaningful data-set will emerge, enabling significant enrichment of our evidence-based understanding of therapeutic processes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing intake to the clinic and beginning therapy

Exclusion Criteria:

* Mental retardation or dementia
* Hebrew Illiteracy
* Adults who are not under their own legal custody
* Not being able to fulfill the questionnaires with minor help

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Overall clinical well-being as measured by the CORE-OM rating scale | up to 3 years follow-up
  The CORE-OM is a short questionnaire that addresses broad psychiatric symptoms including depression, anxiety, well-being, vocational and domestic functioning, social problems, etc.

SECONDARY OUTCOMES:
Hospitalization rates | up to three years of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental Health Center Outpatient clinics, Hod HaSharon, Israel